CLINICAL TRIAL: NCT07296640
Title: A Prospective, Single-Center, Interventional Study to Evaluate the 5-Line Principle of Balanced Intensity Training (BPIT) for Enhancing Physical Performance and Reducing Injury Risk
Brief Title: BPIT 5-Line Pilot: Interventional Study on Strength, HRV & Injury Risk Reduction (n=23)
Acronym: BPIT 5-Line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MMSx Authority Institute for Movement Mechanics & Biomechanics Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPIT-GFFI-2024-001; Other → MMSx Authority (Other Grant/Funding Number: MMSx Authority)
Record Dates: First submitted 2025-11-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPIT 5-Line Training (Experimental): All 23 participants (18 males aged 22-48, 5 females aged 20-33) received BPIT 5-Line Training (3-5 sessions/week, 6 weeks). Intensity progressed via 5 Lines:
  1. Ground-Based, Low Intensity
  2. Knee-Level, Low-Moderate Intensity
  3. Standing, Moderate Intensity
  4. Head-Level, Moderate-High Intensity
  5. Plyometric/High-Impact, High Intensity
  Interventions: Behavioral: BPIT 5-Line Training

INTERVENTIONS:
Behavioral: BPIT 5-Line Training — All 23 participants received BPIT 5-Line Training (3-5 sessions/week, 6 weeks). Intensity progressed via 5 anatomical lines: 1. Ground-Based, Low Intensity; 2. Knee-Level, Low-Moderate; 3. Standing, Moderate; 4. Head-Level, Moderate-High; 5. Plyometric/High-Impact, High Intensity. Sessions 45-60 min, monitored via HRV, pain, fatigue.

SUMMARY:
This prospective, single-center, interventional pilot (n=23) evaluates the 5-Line Principle of Balanced Intensity Training (BPIT) over 6 weeks at GFFI Fitness Academy. Participants (18 males aged 22-48, 5 females aged 20-33) will receive BPIT 5-Line Training (3 sessions/week, 6 weeks). No control group. Conducted July 1 - November 30, 2024.

Progressive intensity via anatomical lines: 1. Ground-Based (Low Intensity); 2. Knee-Level (Low-Moderate); 3. Standing (Moderate); 4. Head-Level (Moderate-High); 5. Plyometric/High-Impact (High). Aims to assess changes in strength, HRV, and injury risk.

DETAILED DESCRIPTION:
STUDY DESIGN: Prospective, single-center, interventional pilot (n=23) with single-group assignment. All participants receive the BPIT 5-Line intervention. Assessments at baseline and Week 6.

INTERVENTION: BPIT 5-Line Training: 3 x 60-minute sessions/week for 6 weeks, progressing across five intensity lines: 1. Ground-Based (Low Intensity, e.g., prone planks); 2. Knee-Level (Low-Moderate, e.g., shoulder press); 3. Standing (Moderate, e.g., half-squat); 4. Head-Level (Moderate-High); 5. Plyometric/High-Impact (High Intensity). Specific exercises detailed in Training Protocol Manual.

OBJECTIVES: Primary - Evaluate BPIT's impact on 1RM strength (e.g., squat, bench press, deadlift) and training-related injury incidence. Secondary - Assess changes in HRV (RMSSD), HRR (bpm in 60s), EMG muscle activation, joint biomechanics (knee valgus, spinal curvature), adherence (% sessions completed), and participant feedback (questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 22-65 years
* Regular fitness trainees (≥2 sessions/week prior)
* Able to provide informed consent
* No recent musculoskeletal injury (past 3 months)

Exclusion Criteria:

* - Cardiovascular disease or uncontrolled hypertension
* Current musculoskeletal injury or surgery (past 6 months)
* Neurological disorders affecting movement
* Pregnancy
* Use of performance-enhancing substances

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in 1RM Strength | 6 weeks
  Change in one-repetition maximum (1RM) strength for key exercises (e.g., squat, bench press) from baseline to week 6. Measured in kilograms (kg) using standard 1RM testing protocol.
  Time Frame: Baseline to Week 6 Unit of Measure: kilograms (kg)
Injury Incidence | Baseline to Week 6
  Number of new musculoskeletal injuries reported during the study period, defined as any complaint requiring medical attention, training modification, or rest exceeding 1 day. Measured as incidence rate per 100 participant-weeks (normalized for exposure in this 23-participant pilot).
  Unit of Measure: injuries per 100 participant-weeks

SECONDARY OUTCOMES:
Change in Heart Rate Variability (HRV) | Week 6
  Change in Heart Rate Variability (RMSSD) from baseline to week 6, measured via 60-second daily monitoring using HRV device/app.
  Time Frame: Baseline to Week 6 Unit of Measure: milliseconds (ms)
Change in Muscle Activation (EMG Amplitude) | Baseline to Week 6
  Change in Electromyography (EMG) amplitude for key muscle groups during specific exercises from baseline to week 6, measured as percentage of maximum voluntary contraction (%MVC) using EMG equipment.
  Time Frame: Baseline to Week 6 Unit of Measure: percentage of maximum voluntary contraction (%MVC)
Change in Joint Biomechanics (Knee Valgus and Spinal Curvature) | Baseline to Week 6
  Change in knee valgus and spinal curvature angles during functional movements from baseline to week 6, measured in degrees via 3D motion analysis or goniometer.
  Time Frame: Baseline to Week 6 Unit of Measure: degrees
Training Adherence | Baseline to Week 6
  Percentage of completed training sessions from baseline to week 6, measured via session logs.
  Time Frame: Baseline to Week 6 Unit of Measure: percentage
Participant Feedback | 6 weeks
  Qualitative feedback from post-study questionnaires, scored on a Likert scale (1-5) for satisfaction and perceived benefit.
  Time Frame: Week 6 Unit of Measure: units on a scale (1-5)
Heart Rate Recovery (HRR) | 6 Weeks
  Change in Heart Rate Recovery (bpm decrease in 60 seconds post-exercise) from baseline to week 6, measured via HR monitor.
  Time Frame: Baseline to Week 6 Unit of Measure: beats per minute (bpm)

CONTACTS AND LOCATIONS:
Locations (1):
- GFFI Fitness Academy, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- See also: Complete Study Documentation Package - BPIT 5-Line Pilot (Protocol, Ethics, Consent, Logs, AE, Report, Closeout) — https://doi.org/10.5281/zenodo.17551763
- Available data/document: Individual Participant Data Set: BPIT-GFFI-2024-001 — https://mmsxauthority.com/BPIT-2024doc.html — De-identified individual participant data (strength, HRV, knee valgus, injury logs) available upon reasonable request to Principal Investigator: Dr. Neeraj Mehta, PhD (info@mmsxauthority.com). All supporting documents (Protocol, Ethics, Consent, Observation Logs, AE Forms, Final Report) uploaded under "Study Documents" tab.

DOCUMENTS (3):
  • Study Protocol (2024-11-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT07296640/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT07296640/SAP_001.pdf
  • Informed Consent Form (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT07296640/ICF_002.pdf